CLINICAL TRIAL: NCT03047148
Title: Immediate Post-operative Outcome After Regional vs. General Anesthesia
Brief Title: Immediate Post-operative Recovery After Regional vs. General Anesthesia
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 2016-01869
Record Dates: First submitted 2017-01-31; First posted 2017-02-08 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Regional Anesthesia: Hospital records from patients who have undergone surgery in regional anesthesia.
  Interventions: Other: Data mining from records
- General Anesthesia: Hospital records from patients who have undergone surgery in General anesthesia.
  Interventions: Other: Data mining from records

INTERVENTIONS:
Other: Data mining from records — The relevant data for this investigation is extracted from the patient records database as well as from the assessment results of the ongoing quality control process that were collected by the nursing staff of the postoperative recovery units.

SUMMARY:
Early post-anesthesia status of patients emerging from surgery encompasses vital respiratory and hemodynamic parameters as well as subjective signs of well-being such as absence of nausea, vomiting and a low pain level. This investigation intends to compare the rate of postoperative complications in the 2 groups from pair matched patient records after regional anesthesia with otherwise similar patients after general anesthesia.

DETAILED DESCRIPTION:
It is still unclear whether the immediate post-operative condition of patients after surgery and anesthesia is dependent on the basic anesthesia technique (General vs. regional anesthesia). The patients' post-anesthesia presentation encompasses vital respiratory and hemodynamic parameters as well as subjective signs of well-being such as absence of nausea, vomiting and a low pain level. By pair matching of patient records after regional anesthesia with otherwise similar patients after general anesthesia (control group), the rate of postoperative complications in the 2 groups will be compared. The results of this investigation will help to answer what is the difference in complication rates and wellbeing of patients depending on their previous anesthesia. The results of this study will Show which basic anesthesia technique has more or less early complications.

ELIGIBILITY:
Inclusion Criteria:

* Records from regional anesthesia cases on adults which have quality control assessment data, plus the same number of matched pairs who had general anesthesia.

Exclusion Criteria:

* Cases with incomplete quality control assessment data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital records from patients after surgery in regional anesthesia that have postoperative quality control data plus a same sized matched pairs control group after general anesthesia.
Sampling Method: Probability Sample
Enrollment: 1880 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Postoperative complications during inhospital stay up to 30 days | 1 March to 30 November 2017
  Number participants who had one or more cardiovascular events up to discharge or 30 days
Postoperative complications during inhospital stay up to 30 days (PONV) - Duration of pain (VAS > 3) episodes in hours; days up to discharge or max. 30 days | 1 March to 30 November 2017
  Number of PONV episodes up to discharge or max. 30 days Duration of PONV episodes in days; hours up to discharge or max. 30 days
Postoperative complications during inhospital stay up to 30 days (pain) | 1 March to 30 November 2017
  Duration of pain (VAS > 3) episodes in hours; days up to discharge or max. 30 days

SECONDARY OUTCOMES:
Length of hospital stay | 1 March to 30 November 2017
  Length of hospital stay in days up to discharge or max. 30 days
Postoperative mortality | 1 March to 30 November 2017
  In-patient postoperative mortality (yes or no up to 30 days)
Total in-hospital costs | 1 March to 30 November 2017
  Absolute amount per case in CHF according financial department report

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Institue of Anesthesiology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
No IPD planned.

REFERENCES:
- [Background] Seims AD, VanHouwelingen L, Mead J, Mao S, Loh A, Sandoval JA, Davidoff AM, Wu J, Wang WC, Fernandez-Pineda I. Operative and Immediate Postoperative Differences Between Traditional Multiport and Reduced Port Laparoscopic Total Splenectomy in Pediatric Patients. J Laparoendosc Adv Surg Tech A. 2017 Feb;27(2):206-210. doi: 10.1089/lap.2016.0309. Epub 2016 Oct 24. PMID 27992299
- [Background] Wood SG, Dabu-Bondoc S, Dai F, Mikhael H, Vadivelu N, Roberts KE. Comparison of immediate postoperative pain after transvaginal versus traditional laparoscopic cholecystectomy. Surg Endosc. 2014 Apr;28(4):1141-5. doi: 10.1007/s00464-013-3294-8. PMID 24232050
- [Background] Neuman MD, Ellenberg SS, Sieber FE, Magaziner JS, Feng R, Carson JL; REGAIN Investigators. Regional versus General Anesthesia for Promoting Independence after Hip Fracture (REGAIN): protocol for a pragmatic, international multicentre trial. BMJ Open. 2016 Nov 15;6(11):e013473. doi: 10.1136/bmjopen-2016-013473. PMID 27852723
- [Background] Moreira CC, Farber A, Kalish JA, Eslami MH, Didato S, Rybin D, Doros G, Siracuse JJ. The effect of anesthesia type on major lower extremity amputation in functionally impaired elderly patients. J Vasc Surg. 2016 Mar;63(3):696-701. doi: 10.1016/j.jvs.2015.09.050. Epub 2015 Nov 6. PMID 26553953